CLINICAL TRIAL: NCT02447887
Title: Phase I/II Study of Ixazomib With Pegylated IFN-alpha 2b (pIFN) in Metastatic Renal Cell Carcinoma (mRCC)
Brief Title: Study of Ixazomib With Pegylated IFN-alpha 2b (pIFN) in Metastatic Renal Cell Carcinoma (mRCC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: IRB study closure facilitated by Investigator
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GU-071; 14-052 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2015-05-06; First posted 2015-05-19 (Estimated); Results first posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Metastatic Renal Cell Carcinoma; RCC
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ixazomib and pegylated IFN alfa - 2b (Experimental): Ixazomib capsules and pegylated IFN alfa 2b injections weekly. Ixazomib will be taken for the last 3 weeks of 28 day cycle. Pegylated IFN alfa 2b injection will be administered weekly, each week of the 28 day cycle.
  Interventions: Drug: Ixazomib; Drug: Pegylated IFN-alpha 2b

INTERVENTIONS:
Drug: Ixazomib — The prescribed administration of ixazomib doses in this study is 1.5-4.0 mg ixazomib weekly for 3 out of 4 weeks in each cycle (1 cycle=28 days).
Drug: Pegylated IFN-alpha 2b — Weekly injection
  Other Names: pIFN - alpha 2b

SUMMARY:
This is a Phase I/II trial of the combination pegylated IFN-alpha 2b with ixazomib in metastatic renal cell carcinoma (mRCC). Researchers believe that by disabling the protein complex NF-kB, which controls the transfer of genetic information; using the study drug Ixazomib, they can promote necrotic cell death of RCC using interferon alpha - 2b. They hypothesize that the combination of ixazomib with IFN will lead to increased necrotic cell death in RCC tumors and consequent clinical benefit to patients.

Patients will receive ixazomib capsules and pegylated IFN alfa 2b injection in this research study. Treatments will be given weekly and 4 weeks of treatment make up one cycle.

ELIGIBILITY:
Inclusion:

1. Male or female patients 18 years or older.
2. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
3. Female patients must be:

   * Postmenopausal for at least 1 year before the screening visit, OR
   * Surgically sterile, OR
   * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
4. Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, or agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
5. Patients must have a diagnosis of a metastatic renal cell carcinoma with a ≥50% clear cell component.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
7. Patients must meet the following clinical laboratory criteria:

   * Absolute neutrophil count (ANC) ≥ 1,000/mm3 and platelet count ≥ 75,000/mm3 and hemoglobin ≥ 9 g/dL. Platelet or red cell transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment.
   * Total bilirubin ≤ 1.5 x the upper limit of the normal range (ULN).
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.
   * Calculated by Cockcroft-Gault creatinine clearance ≥ 30 mL/min (see Section 12.2).
8. Measurable disease by RECIST 1.1.
9. Receipt of at least two line of prior therapy for metastatic RCC.
10. Patients with stable brain metastasis are eligible provided they received definitive therapy (EBRT, gamma knife, surgery) no sooner than 14 days prior to registration and are off all steroids.

Exclusion:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

1. Female patients who are lactating or have a positive serum pregnancy test during the screening period.
2. Failure to have fully recovered (ie, ≤ Grade 1 toxicity) from the reversible effects of prior chemotherapy, radiation therapy or targeted therapy
3. Previous use of interferon, ixazomib or bortezomib.
4. Washout periods for prior therapy are as follows

   * Bevacizumab - last dose must be ≥ 6 weeks prior to day 1 of study treatment.
   * Targeted therapy - last dose must be ≥ 5 half-lives prior to initiation of day 1 of study treatment.
   * Other chemotherapy, immunotherapy, or radiotherapy - Last dose must be ≤ 3 weeks prior to day 1 of study treatment
5. Major surgery within 14 days before enrollment.
6. Radiotherapy within 14 days before enrollment. If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the Ixazomib.
7. Untreated central nervous system involvement.
8. Uncontrolled thyroid disease.
9. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
10. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
11. Systemic treatment, within 14 days before the first dose of Ixazomib, with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
12. Known ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive.
13. Decompensated liver disease (Child-Pugh score >6) or active or past auto-immune hepatitis.
14. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol. In particular, a history of a serous psychiatric illness that might be exacerbated by IFN-α-2b; a history of significant or unstable cardiovascular, hepatic or gastrointestinal disease; a history of autoimmune disease of any kind.
15. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
16. Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing.
17. Evidence of another clinically or radiographically active invasive malignancy OR Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
18. Patient has ≥ Grade 3 peripheral neuropathy, or Grade 2 peripheral neuropathy with pain on clinical examination during the screening period.
19. Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-08-14 (Actual); Primary Completion 2017-04-25 (Actual); Study Completion 2017-04-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ixazomib and Pegylated IFN Alfa - 2b
Started | 3
Completed | 0
Not Completed | 3
Not completed — Study was terminated | 3

BASELINE CHARACTERISTICS:
Population: Only 3 patients total enrolled resulting in IRB closure, deemed a failed trial by the Principal Investigator.The data was never validated and the PI has no intention of having it validated, therefore it cannot be reported.
Arm/Group | Ixazomib and Pegylated IFN Alfa - 2b
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Non-hematologic Toxicity ≥ Grade 3 Per CTCAE v4 Except:
Description: * Grade 3 nausea or Grade 3 vomiting ≤ 72 hours that recovers to grade 0-2 with maximal antiemetic therapy.
  * Grade 3 diarrhea that resolves to grade 0-2 with loperamide or diphenoxylate/atropine within 48 hours.
  * Grade 3 hypercholesterolemia, hypertriglyceridemia, hyperglycemia or hypophosphatemia that resolves to grade 0-2 with medical management.
  * Transient electrolyte abnormalities lasting ≤ 1 week.
Time Frame: Up to week 8
Population: Only 3 patients total enrolled resulting in IRB closure, deemed a failed trial by the Principal Investigator. Data was not validated and PI has no interest in validating the data so it cannot be reported.
Arm/Group | Ixazomib and Pegylated IFN Alfa - 2b
Number analyzed (Participants) | 0

2. Primary Outcome: Thrombocytopenia ≥ Grade 3 Per CTCAE v4
Time Frame: Up to week 8
Population: as for outcome 1
Arm/Group | Ixazomib and Pegylated IFN Alfa - 2b
Number analyzed (Participants) | 0

3. Primary Outcome: Grade 4 Neutropenia Per CTCAE v4; Associated With Fever or Hospitalization for Infection
Time Frame: Up to week 8
Population: as for outcome 1
Arm/Group | Ixazomib and Pegylated IFN Alfa - 2b
Number analyzed (Participants) | 0

4. Primary Outcome: Grade 4 Neutropenia Per CTCAE v4; Lasting Longer Than 5 Days
Time Frame: Up to week 8
Population: as for outcome 1
Arm/Group | Ixazomib and Pegylated IFN Alfa - 2b
Number analyzed (Participants) | 0

5. Primary Outcome: Any Toxicity Felt at the Investigator's Discretion to be Possibly or Probably Related to Ixazomib That Causes the Patient to Miss More Than 1 Dose of Either Ixazomib or pIFN in the First 28 Days.
Time Frame: 28 Days
Population: as for outcome 1
Arm/Group | Ixazomib and Pegylated IFN Alfa - 2b
Number analyzed (Participants) | 0

6. Primary Outcome: Any Unacceptable Toxicity (UT) Defined as Any CTCAE v4 Grade 5 Toxicity, Grade 4 Neuropsychiatric Toxicity or Grade 4 Clinically Significant Non-hematologic Toxicity Thought to be Definitely, Probably or Possibly Related to Study Drug.
Time Frame: 28 Days
Population: as for outcome 1
Arm/Group | Ixazomib and Pegylated IFN Alfa - 2b
Number analyzed (Participants) | 0

7. Primary Outcome: Progression Free Survival Per RECIST 1.1
Time Frame: At week 8
Population: as for outcome 1
Arm/Group | Ixazomib and Pegylated IFN Alfa - 2b
Number analyzed (Participants) | 0

8. Primary Outcome: Progression Free Survuval Per RECIST 1.1
Time Frame: At week 16
Population: as for outcome 1
Arm/Group | Ixazomib and Pegylated IFN Alfa - 2b
Number analyzed (Participants) | 0

9. Secondary Outcome: Overall Response Rate
Time Frame: Week 8
Population: as for outcome 1
Arm/Group | Ixazomib and Pegylated IFN Alfa - 2b
Number analyzed (Participants) | 0

10. Secondary Outcome: Overall Response Rate
Time Frame: Week 16
Population: as for outcome 1
Arm/Group | Ixazomib and Pegylated IFN Alfa - 2b
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: Only 3 patients total enrolled resulting in IRB closure, deemed a failed trial by the Principal Investigator.
Arm/Group | Ixazomib and Pegylated IFN Alfa - 2b
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/87/NCT02447887/Prot_SAP_000.pdf